CLINICAL TRIAL: NCT02998437
Title: A Randomized, Open-label, Parallel-design Study to Evaluate Pharmacokinetic Drug Interactions and Safety After Coadministration of Clarithromycin, Amoxicillin and Ilaprazole
Brief Title: Study to Evaluate Pharmacokinetic Drug Interactions and Safety of Clarithromycin, Amoxicillin and Ilaprazole
Acronym: DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Collaborators: Severance Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IY81149-DI03
Record Dates: First submitted 2016-11-22; First posted 2016-12-20 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Drug Interaction Potentiation
MeSH Terms: interventions — ilaprazole; Clarithromycin; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ilaprazole 10mg (Experimental): Period 1: Ilaprazole 10mg 1 tab.m one a day
  Period 2: Clarithromycin 500mg 1 tab. + Amoxicillin 500mg 2 cap. twice a day, 6 days Ilaprazole 10mg, one a day at the 5 day
  Interventions: Drug: Ilaprazole 10mg
- Clarithromycin 500mg (Active Comparator): Period 1: Clarithromycin 500mg 1 tab. + Amoxicillin 500mg 2 cap., one a day
  Period 2: Ilaprazole 10mg 1 tab., twice a day, 6 days Clarithromycin 500mg 1 tab. + Amoxicillin 500mg 2 cap., one a day at the 5 day
  Interventions: Drug: Clarithromycin 500mg
- Amoxicillin 500mg (Active Comparator): Period 1: Clarithromycin 500mg 1 tab. + Amoxicillin 500mg 2 cap., one a day
  Period 2: Ilaprazole 10mg 1 tab., twice a day, 6 days Clarithromycin 500mg 1 tab. + Amoxicillin 500mg 2 cap., one a day at 5 day
  Interventions: Drug: Amoxicillin 500 Mg

INTERVENTIONS:
Drug: Ilaprazole 10mg — Period 1: Ilaprazole 10mg, one a day, one day Period 2: Ilaprazole 10mg, twice a day, 6 days
  Other Names: Noltec(the brand name)
  Arms: Ilaprazole 10mg
Drug: Clarithromycin 500mg — Period 1: Clarithromycin 500mg 1 tab., twice a day, one day Period 2: Clarithromycin 500mg 1 tab., one a day at 5 day
  Other Names: Klaricid 500mg(the brand name)
  Arms: Clarithromycin 500mg
Drug: Amoxicillin 500 Mg — Period 1: Amoxicillin 500mg 2 cap., one a day, one day Period 2: Amoxicillin 500mg 2 cap., one a day at 5 day
  Other Names: Amoxicillin Cap. 500mg Chongkundang(the brand name)
  Arms: Amoxicillin 500mg

SUMMARY:
This study evaluate the pharmacokinetic drug interaction in Ilaprazole, Clarithromycin, Amoxicillin.

DETAILED DESCRIPTION:
This study evaluate the pharmacokinetic drug interaction and safety in Ilaprazole, Clarithromycin, Amoxicillin.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male adults aged ≥19 years and <50 years at screening
2. Body mass index ≥18.5 and <25

   * Body mass index (kg/m2) = body weight (kg)/[height (m)]2
3. Men who have sexual relationship with women of child bearing potential must give consent to using contraceptive measures (condoms, spermicide, and menstrual cycle control) and avoiding sperm donation during the study and up to 28 days following the last dose of IMP (these contraceptive measures are not required if the male subject or female partner is infertile).
4. Those who voluntarily decided to participate in this study and gave written consent to comply with the requirements after receiving sufficient explanation and fully understanding this study.

Exclusion Criteria:

1. Hypersensitivity or history of clinically significant hypersensitivity to active ingredients or excipients (in particular, Yellow No. 4 (Tartrazine); Yellow No. 5 (Sunset Yellow FCF); macrolide antibiotics such as Clarithromycin and erythromycin; or Penicillins)
2. History of QT prolongation or ventricular arrhythmia (including Torsadedes de pointes)
3. Clinically significant, current or past disorder of hepatobiliary (severe hepatic impairment, etc.), renal (severe renal impairment, etc.), nervous, immune, respiratory, endocrine, blood•tumor, cardiovascular (heart failure, etc.), or psychiatric system
4. History of gastrointestinal disorder (Crohn's disease, ulcer, etc.) or operation (excluding simple appendectomy or herniotomy) that may affect drug absorption
5. Administration of other IMP from other study (including biological comparability test) within 3 months of the first dose of IMP.
6. Whole blood donation within 60 days, or apheresis donation within 30 days before the first dose of IMP.
7. Constant caffeine intake (> 5 cups of coffee/day, > 1250 cc of tea/day, > 1250 cc of cola/day), constant smoking (more than 10 cigarettes/day) or constant alcohol drinking (more than 210 g/week) or inability to refrain from alcohol consumption from 2 days before the first dose of IMP until the end of PK assessment.
8. Consumption of grapefruit-containing food within 7 days before the first dose of IMP
9. History of drug abuse within 1 year before screening, or positive response in urine drug misuse/abuse screening test
10. Use of medicinal products that are expected to or may affect the metabolism of IMP; St. John's wort; or relevant preparations within 30 days of IMP administration
11. Use of following medicinal products within given time period excluding local preparations, which do not have significant systemic absorption, and hormonal contraceptives

    * Prescription drug within 14 days of the first dose of IMP
    * OTC including health supplements and vitamins within 7 days of the first dose of IMP
    * Medicinal products via depot injection or other implantations within 30 days of the first dose of IMP (excluding contraceptives)
    * Drug metabolizing enzyme inducer or inhibitor such as barbiturate within 30 days before the first dose of IMP
12. Stable vital sign measured in sitting position at screening: systolic blood pressure > 150 mmHg or < 90 mmHg, diastolic blood pressure > 100 mmHg or < 50 mmHg, pulse rate > 110 bpm or <40 bpm
13. Following findings at screening

    * Blood total bilirubin > 1.5 x upper limit of normal
    * Blood AST (SGOT), ALT (SGPT) > 1.25 x upper limit of normal
    * MDRD-estimated eGFR < 60 mL/min/1.73m2 eGFR (estimated glomerular filtration rate)(mL/min/1.73m2) = 175 x [serum creatinine (mg/dL)]-1.154 x [age (years)]-0.203
    * Positive serum test (hepatitis B, hepatitis C, HIV, syphilis)
14. Those considered ineligible by the investigator due to other screening results or reasons.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Ilaprazole AUClast(Area Under the plasma concentration-time Curve at the last observed time point) | Predose(0h), after dose 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48h
Ilaprazole Cmax(the maximum serum concentration) | Predose(0h), after dose 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48h
Clarithromycin, Amoxicillin AUClast | Predose(0h), after dose 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48h
Clarithromycin, Amoxicillin Cmax | Predose(0h), after dose 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48h

SECONDARY OUTCOMES:
Ilaprazole AUCinf(Area Under the plasma concentration-time Curve from time zero to infinity) | Predose(0h), after dose 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48h
Ilaprazole Tmax(the time to reach Cmax) | Predose(0h), after dose 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48h
Ilaprazole t1/2(the elimination half-life) | Predose(0h), after dose 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48h
Ilaprazole CL/F(the oral clearance) | Predose(0h), after dose 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48h
Ilaprazole Vd/F(apparent volume of distribution after non-intravenous administration) | Predose(0h), after dose 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48h
Clarithromycin, Amoxicillin AUCinf | Predose(0h), after dose 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48h
Clarithromycin, Amoxicillin Tmax | Predose(0h), after dose 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48h
Clarithromycin, Amoxicillin t1/2 | Predose(0h), after dose 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48h
Clarithromycin, Amoxicillin CL/F | Predose(0h), after dose 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48h
Clarithromycin, Amoxicillin Vd/F | Predose(0h), after dose 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48h

CONTACTS AND LOCATIONS:
Overall Officials: Min MS Park, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Derived] Jin BH, Yoo BW, Park J, Kim JH, Lee JY, Shin JS, Park MS. Pharmacokinetic drug interaction and safety after coadministration of clarithromycin, amoxicillin, and ilaprazole: a randomised, open-label, one-way crossover, two parallel sequences study. Eur J Clin Pharmacol. 2018 Sep;74(9):1149-1157. doi: 10.1007/s00228-018-2489-2. Epub 2018 May 30. PMID 29846770